CLINICAL TRIAL: NCT06911021
Title: 68Ga-FAPI-46 PET/CT for Tumor Fibroblast Imaging to Refine Tumor Assessment and Therapeutic Strategies of Pancreatic Adenocarcinoma
Brief Title: 68Ga-FAPI-46 in Staging of Pancreatic Adenocarcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Giulia Piazza, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI-PANC-2025
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Adenocarcinoma; PET / CT; FAPI; Surgical Oncology; Molecular Imaging
Keywords: Novel imaging in pancreatic cancer; Fibroblast activation protein imaging; Cancer-associated fibroblasts; PET/CT and pancreatic tumor; Tumor microenvironment imaging
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPI-46 PET/CT Imaging Group (Experimental): Single group receiving 68Ga-FAPI-46 PET/CT for diagnostic imaging prior to pancreatic cancer surgery
  Interventions: Diagnostic Test: 68Ga-FAPI-46 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-46 PET/CT — A single-dose intravenous injection of the radiotracer 68Ga-FAPI-46 will be administered to participants. Approximately 60 minutes after injection, a whole-body PET/CT scan will be performed. The scan is designed to detect areas of high fibroblast activation protein (FAP) expression in and around pancreatic tumors, providing high-resolution images of tumor margins and potential spread. The goal is to evaluate whether this imaging method offers more accurate and useful information than standard imaging (MRI and CT) for preoperative staging and surgical planning.

SUMMARY:
This clinical study investigates the use of a new imaging technique called 68Ga-FAPI-46 PET/CT in people with pancreatic ductal adenocarcinoma (PDAC), a type of cancer known for its rapid progression, late diagnosis, and poor survival rate. One of the main challenges with pancreatic cancer is that standard images like MRI and CT, while helpful, are not always able to clearly show how far the cancer has spread or where exactly the tumor ends. This can make surgery and treatment planning more difficult and less precise.

The new image technique being studied, 68Ga-FAPI-46 PET/CT, works by injecting a small and safe amount of a radioactive substance into a vein. This substance travels through the body and attaches to a specific protein called FAP, which is found in large amounts in the tissue that surrounds many pancreatic tumors. By sticking to this protein, the tracer highlights not only the tumor but also the surrounding area that may be affected by the cancer. This results in very detailed images that may show the tumor more clearly than other techniques.

Each participant in the study will receive a single injection of the tracer, and about an hour later they will have the PET/CT scan. The scan itself is quick, painless, and non-invasive, and takes about 20 minutes. A few days later, participants will receive a follow-up phone call to check if they experienced any side effects, though previous studies with over 1,000 people have shown the tracer to be very safe.

The purpose of the study is to find out whether this new technique provides more useful and accurate information than the standard images currently used. It may help better detect the size of the tumor, see if it has spread to other parts of the body, and give doctors a clearer idea of how to plan surgery. This could make it easier to remove the tumor completely and choose the most effective treatment for each patient.

This pilot study is being conducted at Lausanne University Hospital (CHUV) with 20 adult participants over two years. CHUV is the first hospital in Switzerland to offer this kind of scan. If the study is successful, this scan may become a regular part of care for people with pancreatic cancer and could also be used in other cancers in the future.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is one of the most aggressive and deadly types of cancer. It often develops without clear symptoms and is usually diagnosed at a late stage, when treatment options are limited. Even when surgery is possible, the cancer often returns. Current imaging methods like contrast-enhanced CT (ceCT) and MRI are useful tools but have important limitations. They may not clearly show the edges of the tumor, may miss small areas where the cancer has spread, and can be unreliable after chemotherapy, when inflammation can interfere with image interpretation.

This study focuses on a new imaging method called 68Ga-FAPI-46 PET/CT. This technique uses a tracer that attaches to a protein called FAP (fibroblast activation protein), which is found in high amounts in the tissue that supports the growth and spread of pancreatic tumors. These supporting cells, called cancer-associated fibroblasts (CAFs), help the tumor grow, invade nearby tissue, and avoid the immune system. By targeting this protein, the technique can provide highly detailed images of the tumor and the area around it.

Unlike standard PET/CT scans that use sugar-based tracers (such as 18F-FDG), FAPI PET/CT does not rely on the tumor's sugar use to detect it. This is important because many pancreatic tumors do not show up well with FDG scans due to their low activity level. Instead, the FAPI scan focuses on the surrounding tissue that often reacts strongly to the presence of cancer, offering a more complete and accurate picture.

In this prospective study, 20 adult patients with confirmed pancreatic cancer scheduled for surgery will be recruited at Lausanne University Hospital (CHUV). Each participant will receive a single intravenous injection of the 68Ga-FAPI-46 tracer, with the amount based on their body weight. After about 60 minutes, a low-dose PET/CT scan will be performed, taking around 20 minutes. Patients will need to fast for a few hours and drink water before the scan, but no special contrast agents will be used.

After the scan, patients will receive a follow-up call within a few days to check for any side effects. Previous studies have shown that this scan is very well tolerated, with no major side effects reported. Participation in this study will not interfere with any of the patient's normal care or treatment decisions.

The main aim of the study is to compare the results of the FAPI PET/CT scan with those of traditional imaging (CT and MRI) to see which gives better information about the size, shape, and spread of the tumor. Tissue samples collected during surgery will be used to confirm whether what the scan showed matches what is found in real tissue. This will help researchers understand how accurate and useful the scan really is.

Secondary goals include checking whether this technique can show if the cancer has spread to nearby lymph nodes or other organs. It may also help identify areas around the tumor that are more likely to lead to future cancer spread. Knowing this can help in planning surgery and follow-up treatment more precisely.

The study also includes exploratory goals, such as examining the presence of FAP-positive fibroblasts in the removed tissue and how they relate to the PET's results. We hope this will help us learn more about how the cancer behaves and spreads, which could help improve care in the future.

This pilot study will run for about two years. If successful, the results could support the use of 68Ga-FAPI-46 PET/CT as a new standard imaging tool for pancreatic cancer. It may allow for earlier and more accurate diagnosis, better surgical planning, and more personalized treatment decisions. In the future, this imaging technique could also be used for other cancers that involve the same protein, helping more patients benefit from better imaging and care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Karnofsky index ≥80%.
* Operable or operable borderline tumor after neoadjuvant chemotherapy response
* Planned surgical tumor resection.
* SOC imaging (ceCT and MRI) performed as pre-surgery exams.
* Signed informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Claustrophobia.
* Severe renal insufficiency (GFR<30 mL/min/1.73m²).
* Liver enzymes (ALAT, ASAT >5× the upper limit).
* Bilirubin >3× the upper limit.
* Hemoglobin <8 g/dL.
* Absolute neutrophil count <1000/mm³.
* Platelets <75,000/µL.
* Inability to give informed consent or follow study procedures.
* The patient refuses to receive information regarding incidental findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of 68Ga-FAPI-46 PET/CT in Identifying Tumor Size and Spread Before Surgery | From PET/CT scan up to 30 days after surgery
  This outcome will assess how well the 68Ga-FAPI-46 PET/CT scan identifies the size of the primary tumor, its exact borders, and whether it has spread to nearby lymph nodes or other parts of the body, compared to standard imaging methods (MRI and CT). The results will be checked against what is found in the tissue removed during surgery (the gold standard). This will help determine if the new scan provides more precise and useful information for surgical planning and staging.

SECONDARY OUTCOMES:
Detection of Cancer in Lymph Nodes Using 68Ga-FAPI-46 PET/CT | From scan to histological analysis of surgical specimens (up to 30 days after surgery)
  This outcome will evaluate whether the 68Ga-FAPI-46 PET/CT scan can accurately show if the cancer has spread to nearby lymph nodes. The results of the scan will be compared with what is found in the lymph nodes removed during surgery.
Identification of Tumor Infiltration in Surgical Tissue Samples | From scan to histological analysis of surgical specimens (up to 30 days after surgery)
  This outcome will assess if the FAPI PET/CT scan can correctly show where the cancer has invaded tissues that are later removed during surgery. Scan results will be matched with microscopic analysis of those tissues.
Impact of FAPI PET/CT on Surgical and Treatment Planning | From PET to surgery (up to 30 days)
  This outcome will evaluate whether the scan influences how surgery or treatment is planned. The research team will review whether the information from the scan led to changes in the medical team's decisions, such as modifying the surgery or choosing additional treatments.
Safety of 68Ga-FAPI-46 PET/CT | From injection to follow-up call (3-5 days after scan)
  This outcome will track any side effects or safety concerns that occur after the 68Ga-FAPI-46 injection and scan. Patients will be monitored by phone and during follow-up visits, and safety will be evaluated using standard clinical criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is a small, single-center pilot focused on imaging feasibility, and no long-term clinical outcome data will be collected. Additionally, the nature of the data and the limited number of participants may pose a risk of re-identification.